CLINICAL TRIAL: NCT06375733
Title: A Phase Ib/II, Multicenter, Open-label, Single-arm Study to Assess the Safety and Efficacy of GFH009 in Combination With Zanubrutinib in Patients With Relapsed or Refractory Diffuse Large B-cell Lymphoma (DLBCL)
Brief Title: A Study of GFH009 in Combination With Zanubrutinib in Subjects With Relapsed or Refractory DLBCL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genfleet Therapeutics (Shanghai) Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFH009X1202
Record Dates: First submitted 2024-03-05; First posted 2024-04-19 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-03

CONDITIONS: Large B-cell Lymphoma
Keywords: relapsed or refractory diffuse large B-cell lymphoma (DLBCL)
MeSH Terms: conditions — Recurrence; Lymphoma, Large B-Cell, Diffuse | interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1b:GFH009 & Zanubrutinib (Experimental)
  Interventions: Drug: GFH009; Drug: Zanubrutinib
- Phase 2: GFH009 & Zanubrutinib (Experimental)
  Interventions: Drug: GFH009; Drug: Zanubrutinib

INTERVENTIONS:
Drug: GFH009 — administered as an IV infusion at the dose levels 75mg, 60mg, and/or 100mg QW.
  Arms: Phase 1b:GFH009 & Zanubrutinib
Drug: Zanubrutinib — administered at 160mg BID oral; 28-day a cycle until disease progresses.
  Arms: Phase 1b:GFH009 & Zanubrutinib
Drug: GFH009 — the RP2D of GFH009 defined in the preliminary phase 1b trial with the same schedule as in the phase Ib.
  Arms: Phase 2: GFH009 & Zanubrutinib
Drug: Zanubrutinib — administered at 160mg BID oral; 28-day a cycle until disease progresses.
  Arms: Phase 2: GFH009 & Zanubrutinib

SUMMARY:
This is a multicentre, open-label phase Ib/II study. The purpose of the study is to assess the safety and efficacy of GFH009 in combination with Zanubrutinib in patients with relapsed or refractory diffuse large B-cell lymphoma (DLBCL)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Relapsed or refractory diffuse large B-cell lymphoma (DLBCL), including: DLBCL, not specified (NOS), T-cell/histiocyte-rich large B-cell lymphoma (THRLBCL), high-grade B-cell lymphoma, or large B-cell lymphoma transformed from indolent B-cell lymphoma (including but not limited to Richter syndrome, transformed follicular lymphoma, transformed MZL) (2016 WHO classification).
3. Relapse or refractory after receiving 2~4 systemic treatment regimens, at least one of which contains anthracyclines and Rituximab.
4. Must have a measurable lesion.
5. The patient is not suitable to receive stem cell transplantation judged by the investigator.
6. The Eastern Cooperative Oncology Group (ECOG) performance status score (PS) is 0~2.
7. Have adequate organ function, including:

   i. Hematopoietic function: absolute neutrophil count (ANC) ≥1.0×109/L, platelet count (PLT) ≥75×109/L and hemoglobin (Hgb) ≥ 80 g/L.

ii. Liver function: total bilirubin ≤ 1.5 × upper limit of normal (ULN), Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN.

iii. Renal function: Serum creatinine (Cr) ≤ 1.5 × ULN, or serum creatinine clearance ≥ 50 mL/min when Cr > 1.5× ULN.

iv. Coagulation function: International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.

Exclusion Criteria:

1. Primary or secondary central nervous system (CNS) lymphoma.
2. Received chemotherapy, targeted therapy, endocrine therapy, immunotherapy, Chinese patent medicine with anti-tumor effect and other investigational drugs or device therapy within 28 days or 5 half-lives (whichever is shorter), or received therapeutic or palliative radiotherapy within 14 days, or received CAR-T therapy within 12 weeks prior to the administration of the study drugs.
3. Patients with primary resistance to CDK9 or BTK inhibitors.
4. Has a history of organ transplantation or allogeneic stem cell transplantation. Patients who have undergone autologous stem cell transplantation within 6 months.
5. Other malignancies within 2 years prior to study entry, excluding appropriately treated carcinoma in situ of the cervix, focal squamous cell carcinoma of the skin, basal cell carcinoma, prostate cancer not requiring treatment, ductal carcinoma in situ of the breast, and superficial non-muscle-invasive urothelial carcinoma.
6. Have significant diseases of the cardiovascular system or significant acute or chronic infection. History of stroke or intracranial hemorrhage within 6 months prior to enrollment. Presence of significant gastrointestinal disorders. Current clinically significant interstitial lung disease, radiation pneumonitis, or drug-associated pneumonia requiring treatment. Accompanied by other poorly controlled systemic diseases, such as hypertension, diabetes mellitus, etc.
7. Has a history of bleeding disorder or a history of spontaneous bleeding requiring blood transfusion or other medical intervention. Active bleeding within 2 months prior to the first dose.
8. Surgical procedures (excluding needle biopsies) that may affect the administration or study evaluation of this study within 28 days prior to the first dose.
9. Patients who have been treated with prednisone (or equivalent doses of glucocorticoids) at >20 mg/day for anti-tumor purposes within 7 days, or who require long-term use of glucocorticoids for non-anti-tumor therapy.
10. Ongoing medical treatment with a potent inhibitor or inducer of CYP3A is required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: adverse events(AEs) | From Screening (Day -28 to Day-1) to 30 days ±7 days after the last dose, or until the start of a new anti-tumor therapy，assessed up to 32 months
  Incidence of DLT events, incidence and severity of AEs and serious adverse events (SAEs), Electrocardiogram changes
Phase II: ORR | From Screening (Day -28 to Day-1) to 30 days ±7 days after the last dose,or until the start of a new anti-tumor therapy, assessed up to 32 months
  ORR(Objective Response Rate) as assessed by the investigator according to the 2014 Lugano standards

CONTACTS AND LOCATIONS:
Overall Officials: Keshu Zhou, MD, Principal Investigator — Affiliated Cancer Hospital of Zhengzhou University Henan Cancer Hospital
Locations (2):
- China (2):
  - Guangxi Medical University Cancer Hospital&Guangxi Cancer Institute, Nanning
  - Affiliated Cancer Hospital of Zhengzhou University Henan Cancer Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No